CLINICAL TRIAL: NCT05000255
Title: Coping With Covid-19: Loneliness, Self-Efficacy, Social Support and Depression and Anxiety in Patients in Medical Rehabilitation. A Field Study in Geriatrics and Physical Medicine
Brief Title: Coping With Covid-19: Loneliness, Self-Efficacy, Social Support, Depression & Anxiety in Patients in Medical Rehab.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Annette Reichardt, MD (Other)
Collaborators: Jacobs University Bremen gGmbH (Other)
Responsible Party: Sponsor-Investigator, Annette Reichardt, MD, Head of Clinical Trials, Helios Research Center, Helios Research Center
Organization: Helios Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HeliosRC
Record Dates: First submitted 2021-07-25; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Loneliness; Depression, Anxiety; Self Efficacy; Social Support; Covid19; Psychology
Keywords: Loneliness, Depression, Anxiety, Post-COVID, COVID-19, Psych
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: an experimental group comparison is performed. For the first group, a psychological intervention for psychoeducational measures and psychosocial support, was designed according to the recommendations of the DGP - Deutsche Gesellschaft für Pneumologie und Beatmungsmedizin e.V. for the rehabilitation of COVID-19 patients (DGP, 2020). The second intervention was designed after Cacioppo's intervention EASE, for processing loneliness. In this experiment, the psychological interventions will be applied to both groups of patients (non-Covid/post-Covid patients). . Patients who refuse to participate in one of the interventions but nevertheless agree to complete the questionnaires at the measurement time points are treated according to the standards of the complex treatment in early rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1: According to DGP (Experimental): For the first group, a psychological intervention for psychoeducational measures and psychosocial support, was designed according to the recommendations of the DGP - Deutsche Gesellschaft für Pneumologie und Beatmungsmedizin e.V. for the rehabilitation of post-COVID-19 patients (DGP, 2020). The interventions start approximately two days after data collection at T0. The second measurement time point (T1) is scheduled at the time of patient discharge after the interventions have been implemented. Only patients who scored 8 or higher on the Hospital Anxiety and Depression Scale (HADS) at admission will participate in the interventions. This psychological intervention will be applied to both groups of patients (non-Covid/Covid patients)
  Interventions: Behavioral: Intervention 1: According to DGP
- Intervention 2: According to Cacioppo "E.A.S.E." (Active Comparator): The second intervention was designed after Cacioppo's intervention EASE, for processing loneliness. This psychological intervention will be applied to both groups of patients (non-Covid/Covid patients), too. The interventions start approximately two days after data collection at T0. The second measurement time point (T1) is scheduled at the time of patient discharge after the interventions have been implemented. Only patients who scored 8 or higher on the Hospital Anxiety and Depression Scale (HADS) at admission will participate in the interventions.
  Interventions: Behavioral: Intervention 2: According to Cacioppo "E.A.S.E."
- Care as Usual; Standard psychological Support (No Intervention): The patients receive standard care from the psychologists, as is usual in this unit. No intervention is carried out.

INTERVENTIONS:
Behavioral: Intervention 1: According to DGP — The first intervention is designed according to a current recommendation of the Deutsche Pneumologen Gesellschaft e.V. Its approach is resource-oriented, psychoeducational and is expected to have a positive effect on the symptomatology of depression and anxiety in the short and medium term. An additional focus was added to the intervention: planning more physical activity in daily life after discharge. The DPG intervention focuses more on the current state and aims to activate patients' resources in the short and long term. To ensure randomization of study participants, interventions will alternate weekly.
  Arms: Intervention 1: According to DGP
Behavioral: Intervention 2: According to Cacioppo "E.A.S.E." — The second intervention, "E. A. S. E." according to Cacioppo and Patrick (2008), addresses the social action radius of patients (here assuming that loneliness is a predictor of depression). This intervention is about planning social activities against loneliness. Cacioppo's intervention aims to encourage more social activity in the long term.
  Arms: Intervention 2: According to Cacioppo "E.A.S.E."

SUMMARY:
Aim of the study is to investigate possible predictors and factors that may be associated with the development and maintenance of mental and physical health constrains including depression and anxiety symptomatology as well as loneliness in hospitalized post-COVID patients and non-COVID patients in Germany. Furthermore, it will be investigated whether psychological interventions have an effect on anxiety and depression symptomatology, on loneliness values, self-efficacy and perceived social support values. Specifically, the research aim is to examine the relationships between loneliness, self-efficacy, and social support and to address the question of what factors increase the risk of post covid depression/anxiety, and to test the buffering effect of physical and social activities. For this purpose an experimental group comparison will be applied, in which two interventions will be performed on post-COVID patients and non-COVID patients in the unit of Physical Medicine and Geriatrics in Medical Rehabilitation. (PhD Project by Annika Roskoschinski, M.Sc., Psychology, Principal Investigator)

DETAILED DESCRIPTION:
Background: Increased depressive symptoms and anxiety symptoms have been observed in about 23% of all post-COVID patients, also called post-COVID depression (Huang et al., 2021). However, what a) promotes post-COVID depression after the disease and whether it is b) even post-Covid specific has not yet been conclusively understood and will be investigated in this proposed research. The theoretical basis of the proposed work is Cacioppo, Peplau, and Perlman's theory of loneliness, Bandura's self-efficacy theory, and Schwarzer's HAPA model.

Objectives: The aim of the study is to investigate possible predictors and factors that may be associated with the development and maintenance of mental and physical health constrains including depression and anxiety symptomatology as well as loneliness in hospitalized post-COVID patients and non-COVID patients in Germany. Furthermore, it will be investigated whether psychological interventions have an effect on anxiety and depression symptomatology, on loneliness values, self-efficacy and perceived social support values. Specifically, the research aim is to examine the relationships between loneliness, self-efficacy, and social support and to address the question of what factors increase the risk of post covid depression/anxiety, and to test the buffering effect of physical and social activities. For this purpose, a correlational study and an experimental group comparison will be applied, in which two interventions will be performed on post-COVID patients and non-COVID patients. These two data collections will serve as the basis for a later longitudinal study, which is still in the planning stage, as follow-up questions still need to be elaborated. Methods: Around 300 patients should be included in the study. The correlation study at the first measurement point also includes a regression analysis (moderated mediation analysis). Furthermore, an experimental group comparison is performed. For the first group, a psychological intervention for psychoeducational measures and psychosocial support, was designed according to the recommendations of the DGP - Deutsche Gesellschaft für Pneumologie und Beatmungsmedizin e.V. for the rehabilitation of COVID-19 patients (DGP, 2020). The second intervention was designed after Cacioppo's intervention EASE, for processing loneliness. In this experiment, the psychological interventions will be applied to both groups of patients (non-Covid/Covid patients). The interventions start approximately two days after data collection at T0. The second measurement time point (T1) is scheduled at the time of patient discharge after the interventions have been implemented. Only patients who scored 8 or higher on the Hospital Anxiety and Depression Scale (HADS) at admission will participate in the interventions. Patients will be asked to complete the questionnaire again six months after discharge to include a third measurement point and to conduct the aforementioned longitudinal study. Patients who refuse to participate in one of the interventions but nevertheless agree to complete the questionnaires at the measurement time points are treated according to the standards of the complex treatment in early rehabilitation in which a twice psychological contact and screening by means of HADS is obligatory. They form a third group. The following instruments will be used: Items from the UCLA Loneliness Scale (Russel, 1980, German version), the Hospital Anxiety and Depression Scale (Snaith & Zigmond, 2010), Perceived Social Support Questionnaire (F-SozU K-6, Fydrich et al., 2009); SWE - General Self-Efficacy Expectancy Scale (Schwarzer et al., 1999); various self-efficacy instruments, such as staging and Activities Against Loneliness (Lippke, 2007, adapted from Godin & Shepard, 1985). It is expected that self-efficacy and social support play a role as mediator variables and moderator variables and that the symptomatology of depression and anxiety improves after an intervention in COVID and non-COVID patients alike. The findings of this research will contribute to a better understanding of the experience and behavior of patients with and without an infection with COVID-19 in early rehabilitation and identify opportunities for psychological intervention.

The ethics committee of Jacobs University Bremen, where Prof. Dr. Lippke supervises the PhD project, has already approved the research project. Therefore, the project is already in the recruitment phase in order to be able to use data from the third wave from the first quarter of 2021, as this is a special situation in the pandemic and the data would not be reproducible in this way.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years to no upper limit
* patients were diagnosed with COVID-19
* Non-COVID patients with the need to participate in early rehab

Exclusion Criteria:

* a too high language barrier or dyslexia
* patients with intellectual and cognitive impairment (like primary psychiatric illness, e.g., schizophrenia or dementia, if admitted by means of medical history by a physician or if the score achieved in the cognitive screening by means of the mini-mental-state-examination (MMSE) is 23 or below 23 and no improvement of the cognitive performance is to be expected, e.g. because of an incipient dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement with the UCLA Loneliness Scale | approx. 14 days
  Improvement in scores for loneliness: Psychological interventions are expected to improve feelings of loneliness and to decrease loneliness scores.
  The following questionnaire/scale will be used for measurement at the 1st measurement time point and 2nd measurement time point 14 days later for comparison:
  - UCLA Loneliness Scale, German version, short form, 3 Items The lower the scores on the UCLA Loneliness Scale, the better. There is no cut-off Score.
Measurement with the Hospital Anxiety and Depression Scale (HADS) | approx. 14 days
  Improvement in scores for anxiety, and depression: Psychological interventions are expected to improve depression symptomatology and anxiety scores.
  The following questionnaire/scale will be used for measurement at the 1st measurement time point and 2nd measurement time point 14 days later for comparison:
  - HADS - Hospital Anxiety and Depression Scale (HADS-D, German adaptation, 7 items Anxiety, 7 items Depression) A score of 8 or more indicates elevated levels of anxiety and depression. Scores below 8 are targeted by psychological interventions.The cut-off for anxiety and depression is 8 or more.

SECONDARY OUTCOMES:
Measurements with the General Self-Efficacy Expectancy Scale (GSE) | approx. 14 days
  Improvement in scores for self-efficacy: Psychological interventions are expected to increase self-efficacy scores.
  The following questionnaire/scale will be used for measurement at the first measurement time point and 2nd measurement time point 14 days later:
  - General Self-Efficacy Expectancy Scale (GSE), German Version, by Schwarzer, R.
  The higher the values for the above scales, the better. There is no cut-off score.
Measurements of Stage-specific Self-Efficacy, German Version, by Lippke, S. | approx. 14 days
  Improvement of Stage-specific Self-Efficacy:
  Psychological interventions are expected to improve Stage-specific Self-Efficacy.
  The following questionnaire/scale will be used for measurement at the 1st measurement time point and 2nd measurement time point 14 days later:
  - Stage-specific Self-Efficacy, by Lippke, 1 Item, German Version There is no cut-off value.
Measurements of Activities against loneliness, German Version, by Lippke, S. | approx. 14 days
  Improvement of Activities against loneliness:
  Psychological interventions are expected to improve or motivate activities against loneliness.
  The following questionnaire/scale will be used for measurement at the 1st measurement time point and 2nd measurement time point 14 days later:
  - Activities against loneliness, by Lippke, 13 Items, German Version The higher the value for the above scale, the better. There is no cut-off value.
Measurements of Perceived Social Support, (F-SozU K-6), German Short Version, by Fydrich | approx. 14 days
  Improvement in scores for social support:
  Psychological interventions are expected to increase scores of subjectively perceived social support.
  The following questionnaire/scale will be used for measurement at the 1st measurement time point and 2nd measurement time point 14 days later:
  - Perceived Social Support Questionnaire (F-SozU K-6), German Version, by Fydrich (6 Items) The higher the values for the above scales, the better. there is no cut-off value.

OTHER OUTCOMES:
Measurement of loneliness before the COVID-19 pandemic and during the COVID-19 pandemic with prescribed measures (social constraints). | approx. 14 days
  Improving feelings of loneliness during the COVID-19 pandemic.
  * Scale: Feelings of loneliness before and during the pandemic, von Lippke, 2020.
  * 2 items are used
  There is no cut-off value. The lower the scores for loneliness before and during the pandemic, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Study Chair — Jacobs University Bremen gGmbH
Locations (2):
- Germany (2):
  - Helios Klinikum Berlin-Buch GmbH, Berlin
  - Jacobs University Bremen gGmbH, Bremen

IPD SHARING:
Plan to Share IPD: No